CLINICAL TRIAL: NCT05851339
Title: Determinants of Health-related Quality of Life for Patients After Renal Lithotripsy: Percutaneous Nephrolithotomy (PCNL) Versus Retrograde Intrarenal Surgery(RIRS)
Brief Title: Determinants of Health-related Quality of Life for Patients After Renal Lithotripsy: PNL Versus RIRS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Mostafa AbdelRazek, Assistant Professor of Urology, South Valley University
Other Study IDs: SVU/MED/URO016/2.23.4.538
Record Dates: First submitted 2023-05-01; First posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Health Related Quality of Life
Keywords: quality of life , PCNL , RIRS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PCNL: PCNL group applicants will answer SF-36 questionnaire
  Interventions: Other: SF- 36 Questionnaire
- RIRS: RIRS group applicants will answer SF-36 questionnaire
  Interventions: Other: SF- 36 Questionnaire

INTERVENTIONS:
Other: SF- 36 Questionnaire — applicants will fill health related quality of life SF-36 Questionnaire after PCNL or RIRS

SUMMARY:
Percutaneous nephrolithotomy (PNL) and Retrograde intrarenal surgery (RIRS) are well-established procedures for renal stone fragmentation; however, the morbidity, hospitalization, and lost work hours associated with these procedures can negatively affect the health-related quality of life (HRQoL) of the patients [1-3].

The choice of modality is based on the European Association of Urology (EAU) and/or American Urological Association (AUA) guidelines. However, selecting a modality is challenging, considering the advantages and drawbacks of both modalities.

RIRS while minimally invasive, has an inferior stone-free rate compared with PNL; however, PNL requires general anesthesia and longer hospitalization [4]. The need to select the therapeutic modality for urinary lithotripsy based not only on the stone-free rate but also on the subsequent HRQoL of the patient is increasingly recognized [5].

The concept of HRQoL is multidimensional, which includes psychosocial, physical, and emotional factors, as well as patient autonomy, and is applicable to a wide variety of medical conditions [6]. Patients with urolithiasis represent an ideal group for the investigation of HRQoL, considering the disease's high prevalence, non-life-threatening nature, severe symptoms, and high recurrence rate [3]. However, only a few longitudinal studies have investigated HRQoL in patients undergoing lithotripsy for urinary calculi [7]. Several studies have evaluated HRQoL using the Short-Form 36-item survey (SF-36) [3, 7-9].

Hence, this study aims to compare longitudinal HRQoL between PNL and RIRS at four timepoints: before surgery (Bef), on the day of discharge (0 mo), and 1 month (1 mo) and 6 months (6 mo) after surgical intervention, and to further investigate the factors that may significantly affect the HRQoL of these patients

DETAILED DESCRIPTION:
2.4.1- Type of the study: prospective randomized clinical study 2.4. 2- Study Setting: Qena University Hospital 2.4. 3- Study subjects:

1. Inclusion criteria:

   all patients performing PNL or RIRS for renal stones 2-4 cm
2. Exclusion criteria:

   Patients refuse to participate in this study Unfit patients Renal Stones more than 4 cm Renal Stones less than 2 cm
3. Sample Size Calculation:

Not less than 50 patients in each group 2.4.4 -Study tools (in detail, e.g., lab methods, instruments, steps, chemicals, …):

* Medical history
* Complete physical examination.
* Short-Form 36-item survey (SF-36)
* All patents presented was investigated by

  1. Abdominal U.S
  2. Plain X Ray
  3. Non contrast CT
  4. Serum Creatinine
  5. Urine Analysis

ELIGIBILITY:
Inclusion Criteria:

* all patients performing PNL or RIRS for renal stones 2-4 cm

Exclusion Criteria:

* Patients refuse to participate in this study Unfit patients Renal Stones more than 4 cm Renal Stones less than 2 cm

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: all patients presented to our clinics will performing PCNL or RIRS 100 patents in each group
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-07-15 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Determinants of health-related quality of life for patients after renal lithotripsy: PCNL vs RIRS | 2 years
  estimate quality of life patients after PCNL and after RIRS

CONTACTS AND LOCATIONS:
Locations (1):
- South Valley University, Qina, Qena Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No